CLINICAL TRIAL: NCT01954459
Title: Warming up to Sensors: Does Site Warming Improve Continuous Glucose Monitor Performance?
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: unable to complete due to lack of funding
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1306012208; R01DK085618-01 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Continuous glucose sensor; Insupatch
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensor alone (Active Comparator): Glucose sensor site will not have Insupatch
  Interventions: Device: Continuous glucose sensor
- Sensor with Insupatch (Experimental): Glucose sensor site with Insupatch
  Interventions: Device: Insupatch

INTERVENTIONS:
Device: Insupatch — Device which applies local heating at 40 degrees Celsius to the vicinity of the subcutaneous site of glucose sensor.
  Arms: Sensor with Insupatch
Device: Continuous glucose sensor — Glucose sensor inserted without warming patch
  Arms: Sensor alone

SUMMARY:
This study will investigate the effect of wearing a small warming patch, the InsuPatch, at the site of the continuous glucose monitor (CGM), also called a sensor. Specifically, we will be looking to see if using the InsuPatch (IP) improves the accuracy of the continuous glucose monitor.

DETAILED DESCRIPTION:
Hypotheses:

1. Warming of the skin and subcutaneous tissue with the InsuPatch device will improve the accuracy of a CGM as compared to a CGM used alone when both are calibrated with a standard laboratory quality glucose measuring reference standard.
2. Warming of the skin and subcutaneous tissue with the InsuPatch device will reduce the lag time of the CGM, as compared to a CGM used alone when both are calibrated with a standard laboratory quality glucose measuring reference standard.
3. The combination of the InsuPatch device and a CGM will be well-tolerated and not cause skin irritation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least 12 months.
2. Age 8 years to less than 45 years old.
3. Subject understands the study protocol and agree to comply with it.
4. Subject is on insulin pump or injection-based basal-bolus therapy
5. Subject comprehends written English.
6. For females, subject not intending to become pregnant during the study.
7. Informed Consent Form signed by the subject
8. No history of altered skin integrity, poor wound healing, adhesive allergy, or previous infection from sensor wear.
9. Hemoglobin A1C ≤10%

Exclusion Criteria:

1. The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol
2. The presence of any of the following diseases:

   a. Current use of systemic corticosteroids (within the last week) b. Other major illness that in the judgment of the investigator might interfere with the completion of the protocol i. Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
3. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
4. Current or past use of a continuous glucose sensor is not an exclusion criterion.
5. Active skin condition that would affect sensor placement
6. Use of acetaminophen or Vitamin C supplement within the last 7 days
7. Subject is deemed by the Investigator to be unwilling or unable to follow the protocol;
8. Pregnancy A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.

   -

Ages: 8 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Point accuracy of the continuous glucose monitor plus Insupatch (CGM+IP) by mean absolute relative difference (MARD) calculation of sensors with and without IP use. | 4 hours after lunch, 8 hours after breakfast
  Point accuracy of the continuous glucose monitor plus Insupatch (CGM+IP) by mean absolute relative difference (MARD) calculation of sensors with and without IP use, comparing sensor glucose readings and signal data to serum Yellow Springs Instrument (YSI) glucose measurements, with each subject acting as his or her own control.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Michaud, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States